CLINICAL TRIAL: NCT02807649
Title: A 60-Day Clinical Study to Evaluate Nutrilite Ginko Biloba Cistanche Tablets in Relieving the Symptoms of Chronic Fatigue Syndromes Compared to Negative Control
Brief Title: Effect of Ginko and Cistanche Against Fatigue Symptoms
Acronym: GkoCist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Collaborators: Sinphar Pharmaceutical Co., Ltd (Other); Sprim Advanced Life Sciences (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13-SC-4-STL-002
Record Dates: First submitted 2016-01-07; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Mental Fatigue; Fatigue; Chronic Fatigue Syndrome
MeSH Terms: conditions — Mental Fatigue; Fatigue; Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo: Methyl cellulose and dextrose
  Interventions: Dietary Supplement: Placebo Comparator: Placebo
- Low dose (Active Comparator): This blend contains Ginko at 120 mg/day and Cistanche at 300 mg/day
  Interventions: Dietary Supplement: Experimental: Nutrilite® Low dose
- High dose (Active Comparator): This blend contains Ginko at 180 mg/day and Cistanche at 450 mg/day
  Interventions: Dietary Supplement: Experimental: Nutrilite® High dose

INTERVENTIONS:
Dietary Supplement: Experimental: Nutrilite® Low dose — Two tablets consume daily with meal.
  Arms: Low dose
Dietary Supplement: Experimental: Nutrilite® High dose — Two tablets consume daily with meal.
  Arms: High dose
Dietary Supplement: Placebo Comparator: Placebo — Two tablets consume daily with meal.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of Nutrilite® ginkgo biloba cistanche tablets in relieving the symptoms of chronic fatigue syndrome(CFS), the investigators randomly recruit189 subjects with CFS, aged 35-60 yrs. The relief of fatigue and improvement of sexual function are evaluated by World Health Organization Quality Of Life Brief (WHOQoL-Bref), Sexual Life Quality Questionnaire (SLQQ), chronic fatigue syndrome, symptoms of self-assessment at the baseline and the end of intervention. Subjects also underwent a blood test measuring the concentration of biochemical indicators. Cistanche is mainly used to strengthen the renal function, nourish essence and blood in the treatment of lumbar debility, impotence, infertility and muscles weakness, constipation. etc. The study is to test the hypothesis that consecutive 60-day intake of the study tablets can relieve the symptoms of CFS; according to the change of blood biology indicators, the investigators will also evaluate the association between the change of plasma outcome measures and chronic fatigue syndrome.

DETAILED DESCRIPTION:
Chronic fatigue syndrome (CFS) is the common name for a group of significantly debilitating medical conditions characterized by persistent fatigue and other specific symptoms that lasts for a minimum of six months in adults. Symptoms of CFS include malaise after exertion; unrefreshing sleep, physical exhaustion, sore throat, headaches, widespread muscle and joint pain, and depression. The cause of CFS is unclear, but appears to result from a multiple factors. Generally, the onset of CFS is associated with psychological stress, endocrine and immune disorder, genetic factors, and viral infections the diagnostic criteria for CFS modified by Fukuda,etc.in 1994. Currently, there is no one common treatment for CFS. regularly used treatments include the medications which enhance immunity system and nutrition-balanced therapy, Cognitive behavioural therapy (CBT), , local physiotherapy, , and graded exercise therapy(GET).The main purposes of the treatments are to relieve CFS symptoms, improve the psychological condition and social function. According to the U.S. Centers for Disease Control and Prevention (CDC) , CFS will become one of the main diseases that affect human health.

Cistanche, is a desert plants in the family Orobanchaceae. It mainly grows in the sandy pastures of Inner Mongolia, Gansu and Xinjiang Province of China. The plants of the best quality is from Inner Mongolia. According to Traditional Chinese Medical theories, its nature and flavour is sweet, salty, warm, and goes into kidney, large intestine meridians. It is commonly used to invigorate the renal function, nourish essence and blood in the treatment of lumbar debility, impotence, infertility and muscles weakness, and regulates the intestinal tract environment such as dryness, and constipation. A clinical trial showed that Cistanche granules relieved kidney deficiency symptoms in 86.7% of the chronic fatigue syndrome patients, demonstrated a significant difference comparing post-intervention to baseline (P <0.01).

Ginko As recorded in the Yuan Herbal Classic by Lulu Zhang Feng in Qing Dynasty, ginkgo has functions of reducing phlegm, detoxification, insect killing, could cure scabies and gangrene tumors, acute mastitis ulceration disease, dental caries, infantile diarrhea, leukorrhea with reddish discharge, chronic stranguria with turbid discharge, emission enuresis disease.

In addition, ginkgo can inhibit various types of pathogenic bacteria. A clinical study (conducted by Wuhan Military General Hospital) of over 100 subjects with high cholesterol showed that ginkgo extract (guanxin ketones) has antihypertensive effect.

Germany, United Kingdom, France, USA and South Korea also used ginkgo leaves to produce drugs for treating cardiovascular and cerebrovascular diseases.

Ginkgo root, containing ginkgo lactone C, M, A, B, is sweet, warm, plain and nontoxic, and can be used to treat leucorrhea disease and emission.

A study about late Alzheimer disease found that ginkgo can improve vascular patency, thus has notable effect in anti-aging of brain function in elderly people, and enhancing memories.

Subjects with ginkgo juice supplement showed significant improvement in memory, attention and complex movements compared to the control group, patients who take ginkgo juice have significantly improved.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed as CFS by general practitioner and at least have four symptoms:

memory loss or lack of concentration, muscle pain, sleep disturbances, continuous discomfort after labor; Or be diagnosed as CFS according to the clinical diagnosis 30-60 days before screening;

* Have normal electrocardiograms (ECG) and blood pressure during quiet respiration and during exercises.
* Be willing to use reliable contraception methods during the study period (only for volunteers with fertility).
* Agree not to take any medication, supplement or nutrition with promoting function to exercise capacity;
* Be willing to comply with all the requirements and procedures of the study;
* Agree to sign the informed consent form;
* Fully understand the nature, objective and the potential risks and side effects of the study.

Exclusion Criteria:

* BMI≧28；
* Female on menopausal；
* Have participated in similar clinical trials within 6 months before the screening;
* Currently taking medicines for cardiovascular or metabolic disease ;
* Have flu/symptoms of viral infection within three months before the first visit;
* Have history of or be diagnosed of any of the following diseases that may affect the study results: gastrointestinal disorders, hepatopathy, nephropathy, endocrine disease, blood disorders, respiratory and cardiovascular diseases;
* Current or previous alcohol abuser, currently taking or took illicit drugs, substance or over the counter prescription drugs which promote athletic performance;
* Subject with iron-deficiency anemia, diabetes mellitus, epilepsy, bleeding tendency or Coagulation disorders;
* Currently suffering from any gastrointestinal disorders or skeletal muscle dysfunction, including but not limited to: irritable bowel syndrome, colitis, ulcerative colitis, celiac disease, osteoporosis or arthritis;
* Currently having or had any medical or nutritious therapies, including taking protein supplements or nutrients that promote exercise capacity within 3 months before screening;
* Have lost or gained weight over 5 kilograms within 3 months before screening;
* Had hospitalizations within 3 months before screening;
* According to investigator's judgement, current frequent users of drugs which may affect the electrolyte balance or hydration.
* Pregnant or nursing female, as determined by a questionnaire.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Net change in the score of World Health Organization Quality of Life survey before and after intervention | 60 days

SECONDARY OUTCOMES:
Net change in the score of Chalder fatigue scale survey before and after intervention | 60 days
Net change in the score of Chalder fatigue self assessment survey before and after intervention | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Shuguang Li, PhD, Principal Investigator — Fudan University, Department of Nutrition and Food Hygiene

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Li Y, He DJ, Jiang ZL, Wu YQ and al. Studies on Emotional characteristics of individuals with chronic fatigue syndrome. China Journal of rehabilitation medicine, 2006, 21(3):218-220
- [Background] 2. Zhang J. Clinical study on behavior intervention in chronic fatigue syndrome. Liaoning Journal of Traditional Chinese Medicine, 2009, 36(8):1338-1340.
- [Background] Fukuda K, Straus SE, Hickie I, Sharpe MC, Dobbins JG, Komaroff A. The chronic fatigue syndrome: a comprehensive approach to its definition and study. International Chronic Fatigue Syndrome Study Group. Ann Intern Med. 1994 Dec 15;121(12):953-9. doi: 10.7326/0003-4819-121-12-199412150-00009. PMID 7978722
- [Background] 4. Shen XH, Zheng L, Zhu WR, Xu JZ, Chen JX and al. Clinical effect observation of Cistanch Yishen granule in the treatment of kidney deficiency type of chronic fatigue syndrome. China Pharmacy, 2008, 19(18):1416-1418.
- [Background] 5. Jean Carper.Magical Food.Beijing: Xinhua Publishing
- [Background] Dou GX. Diet Guide, 1981, Jiangsu Sci and Tech Publishing.
- [Derived] Kan J, Cheng J, Hu C, Chen L, Liu S, Venzon D, Murray M, Li S, Du J. A Botanical Product Containing Cistanche and Ginkgo Extracts Potentially Improves Chronic Fatigue Syndrome Symptoms in Adults: A Randomized, Double-Blind, and Placebo-Controlled Study. Front Nutr. 2021 Nov 26;8:658630. doi: 10.3389/fnut.2021.658630. eCollection 2021. PMID 34901100